CLINICAL TRIAL: NCT06128720
Title: A Randomized, Sham Controlled, Masked Phase II Study to Evaluate the Neuroprotective Effect of Hyperbaric Oxygen Therapy on Optic Neuropathy
Brief Title: Hyperbaric Oxygen Therapy for Optic Neuropathies
Acronym: HBOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59547
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Optic Neuropathy; Glaucoma
MeSH Terms: conditions — Optic Nerve Diseases; Glaucoma | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Open Label (Experimental): Participants will get Hyperbaric oxygen therapy for 20 days to determine best methods for full trial.
  Interventions: Device: Hyperbaric Oxygen
- Active Hyperbaric Oxygen (Experimental): Participants will get Hyperbaric oxygen therapy for 20 days.
  Interventions: Device: Hyperbaric Oxygen
- Sham Hyperbaric Oxygen (Placebo Comparator): Participants will get a Sham Hyperbaric oxygen therapy for 20 days
  Interventions: Device: Sham Hyperbaric Oxygen

INTERVENTIONS:
Device: Hyperbaric Oxygen — Participant will undergo 60 minutes of Hyperbaric oxygen at 1.5ATA while breathing 100% oxygen
  Arms: Active Hyperbaric Oxygen; Open Label
Device: Sham Hyperbaric Oxygen — Participant will undergo 60 minutes of Sham Hyperbaric Oxygen at atmospheric pressure while breathing room air.
  Arms: Sham Hyperbaric Oxygen

SUMMARY:
The purpose of the study is to evaluate the neuroprotective efficacy of hyperbaric oxygen for the treatment in patients with optic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to join the study (all eligibility criteria must be met at the screening and baseline visits unless otherwise noted):
* Participant must be at least 18.
* Participant must has the ability to comply with the requirements of the study and complete the schedule of events (SOE).
* Participant's with clinical evidence of optic neuropathy.
* Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.

Exclusion Criteria:

* Participant is unable to comply with study procedures or follow-up visits.
* Participant has evidence of corneal opacification or lack of optical clarity.
* Participant is currently participating in or has within the last 3 months participated in any other clinical trial of a drug by ocular (if in the study eye) or systemic administration.
* Participant is pregnant or lactating.
* Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments.
* Children and comatose patients.
* Participant abusing drugs or alcohol.
* Prior treatment with hyperbaric oxygen within the last 6 months.
* Participant with claustrophobia or that cannot decompress properly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Field- Mean Deviation | Baseline through 6 months
  Humphrey visual field testing with standard MD output
Change in Visual Field- Visual Field Index | Baseline through 6 months
  Humphrey visual field testing with standard VFI output

SECONDARY OUTCOMES:
Change in Average Thickness Ganglion Cell Complex on Optical Coherence Tomography | Baseline through 6 months
  OCT testing with standard GCC output
Change in Average Thickness Retinal Nerve Fiber Layer on Optical Coherence Tomography | Baseline through 6 months
  OCT testing with standard RNFL output

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD PhD, Study Chair — Stanford University
Locations (1):
- Byers Eye Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No